CLINICAL TRIAL: NCT06036290
Title: Study of the Association Between the Discordance in the Evaluation of Suicidal Intentionality Between Parents and Adolescents After a Suicide Attempt in Adolescence and the Evolution of the Suicidal Crisis at 3 Months: a Mixed Study
Brief Title: Discordance in the Evaluation of Suicidal Intent Between Parents and Adolescents in Adolescence and Evolution of the Suicidal Crisis : a Mixed Study
Acronym: discord-Ados
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2023 SIBUT
Record Dates: First submitted 2023-08-08; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Suicidal Intention; Suicide, Attempted; Parent-Child Relations
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this mixed-methods study is to describe the association between the level of parent/adolescent discordance in the assessment of the adolescent's level of suicidal intentionality after a suicid attempt and the evolution of the suicidal crisis by assessing the evolution of the adolescent's suicidal intentionality between T0 and 3 months.

The main questions it aims to answer are:

* To show the association between the level of parent/adolescent discordance in the assessment of the adolescent's level of suicidal intent after a suicid attempt and various markers of the evolution of the suicidal crisis at 3 months.
* Explore the experience of adolescents and their parents regarding the elements they consider relevant in assessing the adolescent's suicidal intent.

Participants will be asked to complete various self- and hetero-questionnaires at T0 and T3

DETAILED DESCRIPTION:
Mixed quantitative and qualitative descriptive observational study. Participants will be included at the various sites by the investigators attached to the three inclusion sites.

Primary outcome

Difference in adolescents' level of suicidal intent between T0 and 3 months. All measurements are with a Visual Analogue Scale (VAS) graded from 0 to 10.

Secondary outcomes Quantitative study

* Total number of new suicidal crisis-related visits to the emergency department and/or the child psychiatry emergency and mobile team at 3 months.
* Total number of suicidal recurrences at 3 months.
* Total number of full-time inpatient stays in MCO and/or psychiatry related to suicidal crisis at 3 months.
* Total length of stay in full-time inpatient care (MCO and/or psychiatry) related to suicidal crisis at 3 months.
* Proportion of the number of days of absence out of the total number of school days at 3 months.
* Proportion of number of child psychiatric consultations honored out of total number of scheduled consultations at 3 months.
* Proportion of the number of psychological consultations honored out of the total number of consultations scheduled for 3 months.
* Total score on FACES IV self-assessment scale of family functioning.
* Gender, age, urban or rural environment, family organization (union, single parent, other situations) and parents' socio-professional category.
* i) Presence of a family psychiatric history; ii) Presence of a family suicide history; iii) Presence of a family history of TS; iv) Presence of a personal history of TS; v) Presence of a personal history of psychological or psychiatric follow-up; vi) Presence of a personal history of self-harm; vii) Type of TS and viii) Type of ICD-10 diagnosis made during the child psychiatric assessment.
* Difference in adolescents' level of suicidal intentionality measured using a Visual Analog Scale at: i) T0 (measurement of level 1 week prior to TS, level at time of TS, level at time of assessment) and ii) T3 months.
* Difference in level of parent/adolescent suicidal intentionality measured at T0 and T3 months using the VAS.

Qualitative study

* Obtaining a thematic grid describing the experience of adolescents and their parents regarding the elements they consider relevant in assessing the adolescent's suicidal intent.
* Obtained a thematic grid describing the experience of adolescents and their parents regarding their mutual understanding of the suicidal crisis experienced by the adolescent.

The study is descriptive, and qualitative for a subsample of participants.

- Hetero-questionnaire 1: Hetero-questionnaire 1 collects socio-familial and clinical data at T0. Data are collected by the investigator on the day of inclusion in the study. The main elements collected are

* Patient's gender
* Patient's age
* rural or urban environment
* Family organization
* Parents' socio-professional category
* Family history of suicide
* Presence of a family history of suicidal attempt
* Presence of a personal history of suicidal attempt
* Personal history of psychological or psychiatric treatment
* Personal history of self-mutilation
* Type of suicidal attempt
* ICD-10 diagnosis made during child psychiatric assessment
* Hetero-questionnaire 2:

Hetero-questionnaire 2 is used to collect declarative data on progress at T3months. Data are collected by an authorized member of the study, by videoconference. Parents will be informed of the need for the child to be alone at the time of the interview, in a quiet, dedicated room. The main data collected are

* The total number of new consultations with the emergency department and/or the mobile child psychiatry team in connection with the suicidal crisis at 3 months.
* Total number of suicidal attempts recurrences
* Total number of full-time hospital stays related to the suicidal crisis.
* Total length of stay in full-time hospitalization related to suicidal crisis.
* Number of days of absence as a proportion of school days
* The proportion of the number of child psychiatric consultations honored out of the total number of scheduled consultations
* The proportion of the number of psychological consultations honored out of the number of scheduled consultations
* Auto-questionnaire FACES IV
* Semi-structured interviews Semi-structured interviews are specifically designed to explore the various themes announced. An interview guide is drawn up by the research group, made up of specialists in adolescent psychiatry and qualitative methods. The guide is not fixed, contains "starter" questions and can be modulated as the research progresses. The researcher has in mind a list of themes that must necessarily be addressed, but the discussion remains very open, in order to enter the subject's internal world. The subject acts as an expert, and may bring up one or more themes that the researcher hadn't thought of, depending on his or her concerns and interests.

Two interviews are conducted, one with the adolescent, the other with his or her parents. The interviews with the patients and their parents explore the parents' and the adolescent's experience of the suicidal crisis, family relationships and how they evolved during the crisis.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents:
* aged 11 to 17
* admitted to a pediatric or adult emergency department following a suicide attempt
* proficient in spoken French
* not opposed to participation in the research
* accompanied by at least one parent who is not opposed to the adolescent's participation in the research.
* Parents:
* 18 years of age or older
* parent or guardian of an adolescent admitted to a pediatric or adult emergency department following a suicide attempt
* fluent in spoken French
* not opposed to participation in the research

Exclusion Criteria:

* present a decompensated somatic or psychiatric pathology or a vigilance disorder
* refusal to participate in the research

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents: aged 11 to 17, admitted to a pediatric or adult emergency department following a suicide attempt.
  Parents: 18 years of age or older, parent or guardian of an adolescent admitted to a pediatric or adult emergency department following a suicide attempt.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-05-27 (Estimated); Study Completion 2025-05-27 (Estimated)

PRIMARY OUTCOMES:
Difference in adolescents' level of suicidal intent | 3 months
  Difference in adolescents' level of suicidal intent between T0 and 3 months. All measurements are based on a Visual Analogue Scale (VAS) graduated from 0 to 10.

SECONDARY OUTCOMES:
Association between the level of parent/adolescent discordance in the assessment of the adolescent's level of suicidal intent after a suicidal attempt and various indicators of the evolution of the suicidal crisis at 3 months. | 3 months
  * Total number of new emergency room and/or child psychiatry team consultations related to suicidal crisis at 3 months.
  * Total number of suicidal recurrences reported at 3 months.
  * Total number of full-time inpatient hospital stays or psychiatry related to the suicidal crisis at 3 months.
  * Total length of stay in full-time in-patient care in the hospital, and/or psychiatry, related to the suicidal crisis at 3 months.
  * Proportion of the number of days of absence out of the total number of school days at 3 months.
  * Proportion of number of child psychiatric consultations honored out of total number of scheduled consultations at 3 months.
  * Proportion of the number of psychological consultations honored out of the total number of consultations scheduled at 3 months
association between the level of parent/adolescent discordance in assessing the adolescent's level of suicidal intent after a suicid attempt and the degree of family cohesion | 1 week
  Total score on FACES IV self-assessment scale of family functioning.
socio-familial factors associated with a high level of parent/adolescent discordance in assessing the adolescent's level of suicidal intentionality after a suicidal act. | 1 week
  Gender, age, urban or rural environment, family organization (union, single parent, other other situations) and parents' socio-professional category.
clinical factors associated with a high level of parent/adolescent discordance in assessing the adolescent's level of suicidal intent after a suicide attempt. | 1 week
  i) presence of a family psychiatric history; ii) presence of a family suicide history; iii) presence of a family history of suicide attempt; iv) presence of a personal history of suicide attempt; v) presence of a personal history of psychological or psychiatric follow-up; vi) presence of a personal history of self-harm; vii) type of suicide attempt and viii) type of ICD-10 diagnosis made during the child psychiatric evaluation.
evolution of the level of parent/adolescent discordance on the evaluation of the adolescent's level of suicidal intent after a suicide attempt at 0 and 3 months | 3 months
  Difference in the level suicidal intent of adolescents measured with a Visual Analog Scale at scale at: i) T0 (measurement of level 1 week prior to suicidal event, level at time of suicidal event level at the time of TS, level at the time of assessment) and ii) T3 months
Explore the experience of adolescents and their parents regarding the elements they consider relevant in assessing the adolescent's suicidal intent. | 1 month
  Obtained a thematic grid describing the experience of adolescents and their parents with regard to the elements they consider relevant in assessing the adolescent's suicidal intent.
Explore the experience of adolescents and their parents in terms of their mutual understanding of the suicidal crisis experienced by the adolescent. | 1 month
  Obtaining a thematic grid describing the experience of adolescents and their parents in terms of their mutual understanding of the suicidal crisis experienced by the adolescent.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No